CLINICAL TRIAL: NCT01702181
Title: A Multiple-Dose (0.3%, 1%, and 3% [w/w]), Randomized, Blinded, Vehicle- and Active Comparator-Controlled, Sequential Dose Cohorts, Multi-Center Trial to Assess the Safety, Pharmacokinetics, and Proof-of-Concept Efficacy of Topical OPA 15406 Ointment, Applied Twice Daily for 28 Days, in Adult Subjects With Atopic Dermatitis
Brief Title: A Safety Study to Evaluate the Use and Effectiveness of a Topical Ointment to Treat Adults With Atopic Dermatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 271-12-204
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis, Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — difamilast; Tacrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Matching placebo.
  Interventions: Drug: Placebo
- Tacrolimus (Active Comparator): Tacrolimus 0.1% ointment twice daily for 28 days.
  Interventions: Drug: Tacrolimus
- OPA-15406 (Experimental)
  Interventions: Drug: OPA-15406

INTERVENTIONS:
Drug: OPA-15406 — 0.3%, 1%, or 3% OPA-15406 topical ointment, applied twice daily for 28 days
  Arms: OPA-15406
Drug: Tacrolimus — 0.1% concentration of tacrolimus.
  Other Names: Protopic
  Arms: Tacrolimus
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics and safety of OPA-15406 in adult subjects with atopic dermatitis

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects 18-65 years of age
* Diagnosis of atopic dermatitis (AD)
* AD affecting at least 5% of total Body Surface Area (BSA) for Part 1 and at least 10% BSA for Part 2, not including face, neck, and head
* Have had a positive but inadequate response to one or more treatment course of standard AD therapy including topical steroids, UV light A, narrowband UV B, and UV light B.

Exclusion Criteria:

-Use of systemic or topical therapy for contact or atopic dermatitis within 30 days of screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2012-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects with AEs, SAEs, and % of clinically relevant changes from baseline in Draize Scale, physical examinations, vital signs, laboratory assessments, and electrocardiograms. | 28 days
Measurement of drug levels in the blood of treated patients | 28 days

SECONDARY OUTCOMES:
Investigator's Global Assessment (IGA) of Disease Severity at Week 4 | 28 Days

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Mobile, Alabama
  - Hot Springs, Arizona
  - Irvine, California
  - Orange Park, Florida
  - Tampa, Florida
  - Carmel, Indiana
  - Berlin, New Jersey
  - High Point, North Carolina
  - Portland, Oregon
  - College Station, Texas
  - Dallas, Texas
  - San Antonio, Texas